CLINICAL TRIAL: NCT05503134
Title: Killer Cells Against Relapsed/Refractory Myeloid Acute Leukemia (KARMA): a Clinical Trial Evaluating the Safety and Efficacy of Expanded, Universal Donor Natural Killer Cells for Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Safety and Efficacy of Expanded, Universal Donor Natural Killer Cells for Relapsed/Refractory AML
Acronym: KARMA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KARMA
Record Dates: First submitted 2022-02-14; First posted 2022-08-16 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Fludarabine 30 mg/m2/day (day -6 to day -2) and Cytarabine 2000 mg/ m2/day (days -6 to day -2)
  Six doses of universal donor IL-21 expanded NK cells (UD-NK) given thrice weekly for two weeks starting on day 0. Days may vary and NK cells can be given from days 0 to 21. Patients may receive up to 2 cycles of fludarabine/cytarabine (FLA) + NK cells (up to 12 NK cell infusions) if they do not achieve CR after cycle 1 or if necessary to bridge to transplant.
  Interventions: Biological: Universal Donor Natural Killer Cells

INTERVENTIONS:
Biological: Universal Donor Natural Killer Cells — Six doses of UD-NK cells will be given thrice weekly for two weeks for up to 2 cycles of treatment

SUMMARY:
This is a phase I/II dose escalation study designed to determine the safety and estimate the efficacy of UD-NK cells combined with FLA chemotherapy in patients age 1-24.99 with relapsed or refractory acute myeloid leukemia.

PRIMARY OBJECTIVE:

I. To determine the safety and recommended phase II dose of adoptive NK cell therapy using UD-NK cells in pediatric and young adult patients with relapsed/refractory AML.

SECONDARY OBJECTIVES:

I. To estimate the efficacy of UD- NK cells with FLA chemotherapy in pediatric and young adult patients with relapsed/refractory AML.

EXPLORATORY OBJECTIVES:

I. To determine the immunophenotype and function of UD-NK cells

II. To characterize in vivo expansion of UD-NK cells

III. To determine the persistence of UD-NK cells

Six doses of universal donor mbIL-21 expanded NK cells (UD-NK) given thrice weekly for two weeks. Days may vary and NK cells can be given from days 0 to 21. Patients may receive up to 2 cycles of fludarabine/cytarabine (FLA) + NK cells (up to 12 NK cell infusions) if they do not achieve CR after cycle 1 or if necessary to bridge to transplant.

DETAILED DESCRIPTION:
The treatment plan consists of Fludarabine/Cytarabine chemotherapy followed by six doses of universal donor mbIL-21 expanded NK cells (UD-NK) given thrice weekly for two weeks. Days may vary and NK cells can be given from days 0 to 21. Patients may receive up to 2 cycles of fludarabine/cytarabine (FLA) + NK cells (up to 12 NK cell infusions) if they do not achieve CR after cycle 1 or if necessary to bridge to transplant.

In this study the first NK cell infusion is referred as day zero (D0), treatment plan activities prior or after D0 are denominated as day minus (D-) or day plus (D+).

FLA will be give as follows: Fludarabine 30 mg/m2/day (day -6 to day -2) and Cytarabine 2000 mg/ m2/day (days -6 to day -2)

Six doses of UD-NK cells will be given thrice weekly for two weeks beginning day 0. NK cell administration schedule may vary and doses may be given from day 0 to 21. A minimum of 2 days between NK cell doses is required. Patients must meet eligibility criteria for NK cell infusion as described in the protocol.

Patients will be eligible to receive a second cycle of chemotherapy for the following reasons:

1. <CR after cycle 1
2. Additional cycle is needed to bridge the patient to HSCT

Criteria to begin Cycle 2:

1. ≥28 days since the first NK Cell infusion
2. ≥2 days since the last NK Cell infusion in cycle 1
3. Bone marrow evaluation after cycle 1 complete
4. It is suggested but not required for ANC > 500/uL AND platelets >50,000/uL prior to beginning cycle 2
5. Prior treatment related toxicities must have resolved to ≤ Grade 2

NK Cell Dose Levels:

1. Dose level 1: 1.00x10^7 NK cell/kg (±20%) each dose for 6 doses per cycle
2. Dose level 2: 3.00x10^7 NK cell/kg (±20%) each dose for 6 doses per cycle
3. Dose level 3: 1.00x10^8 NK cell/kg (±20%) each dose for 6 doses per cycle

The NK dose will be calculated based on actual body weight. Dose escalation will proceed according to the study design outlined in Section 9.1 to determine the MTD. Once a patient is enrolled at a dose level, the dose will remain at the enrolled dose level for all subsequent NK cell infusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or primary refractory AML, including:

  * Patients with relapsed AML (Any patient in first or subsequent relapse are eligible. Patients with relapse after HSCT are eligible)
  * Primary refractory AML defined as failure to achieve a complete response after 2 cycles of induction chemotherapy, including persistent MRD positivity
  * Patients with isolated CNS or extramedullary disease are eligible Note: a response monitoring plan must be developed a priori for subjects with extramedullary disease
* Patient age 1-24.99 years old
* Negative serum test to rule out pregnancy within 2 weeks prior to enrollment in females of childbearing potential

  o Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator for 6 months after the last dose of chemotherapy and/or NK cell infusion
* Negative serology for human immunodeficiency virus (HIV)
* Both males and females and members of all races and ethnic groups are eligible
* Organ function requirements:

  * Renal function: Creatinine ≤ 2 mg/dl OR creatinine clearance > 60 ml/min/1.73m2.
  * Liver function: Total bilirubin ≤ 2 mg/dl (unless Gilbert's syndrome), AST and ALT ≤ 5 times the upper limit of normal (unless related to leukemic involvement). Upper limit of normal should be determined by the institutional defined normal laboratory range.
  * Cardiac function: left ventricular ejection fraction ≥ 40% or shortening fraction ≥20%. May be eligible after cardiology clearance if qualitatively normal function or repeat measures are normal.
  * CNS: Patients with seizure disorder may be eligible if seizures well controlled
* All prior treatment related non-hematologic toxicities must have resolved to ≤ Grade 2 prior to enrollment unless granted approval by study PI and/or Co-Is.
* All patients and/or their legal guardians must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* AML directed therapies in the 2 weeks prior to beginning treatment on this protocol (except for hydroxyurea)

  o Note: There is no waiting period required for patients having received intrathecal cytarabine, methotrexate and/or hydrocortisone
* Patients on immunosuppressive therapy

  o Patients must be off of all systemic immunosuppressive therapy for at least 2 weeks prior to enrollment with no evidence of recurrent GVHD
* Patients with a history of donor lymphocyte infusion or cellular therapy within the last 30 days are not eligible for this study
* Allogeneic SCT < 3 months prior to study enrollment
* Any comorbidities that in the opinion of the investigator will preclude receiving study therapy
* Performance status: Karnofsky or Lansky Performance Scale (PS) < 50
* Uncontrolled infection, defined as an infection which has not resolved or does not show evidence of significant resolution after initiating appropriate therapy

  o Asymptomatic viremia such as CMV, HPV, BK virus, HCV, etc. is NOT considered as an exclusion criterion
* Uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease
* History of autoimmune disease
* Active GVHD at the time of enrollment
* Patients with a history of adoptive cell therapy are excluded unless at least 30 days from infusion and with evidence of recovery of normal hematopoiesis (ANC ≥ 500/μL, platelet count ≥ 50,000/μL).

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 56 days after the first NK cell infusion
Rate of dose limiting toxicities | Up to 56 days after the first NK cell infusion

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) negative response rate by flow cytometry | At the end of Cycle 1 and Cycle 2 (each cycle is 28 days)
CR rate after first cycle | At the end of Cycle 1 (each cycle is 28 days)
Relapse free survival and overall survival | 1 year
Median time to neutrophil and platelet count recovery | 1 year
Median duration of remission for patients who do not go onto transplant | 1 year
Incidence of infectious complications | 1 year
Percentage of patients receiving this regimen who are rendered transplant-eligible | 1 year

OTHER OUTCOMES:
Immunophenotype of UD-NK cells | Weekly samples from day 0 to day +28 after the first NK cell infusion for each cycle (each cycle is 28 days)
  Immunophenotyping by flow cytometry and CyTOF.
Function of UD-NK Cells | Day 0 of the first cycle
  Cytokine secretion and cytotoxicity of UD-NK cells cultured with patient leukemia samples
Expansion/persistence of UD-NK cells after infusion | Weekly samples from day 0 to day +28 after the first NK cell infusion for each cycle (each cycle is 28 days)
  Peripheral blood will be obtained before therapy, during the NK cell treatment period, and after NK cell treatment to evaluate for UD-NK cell expansion and persistence. UD-NK cells will be identified by chimerism assay. Chimerism may be determined by flow cytometry using haplotype-specific antibodies, short tandem repeat polymorphisms, or when there is a sex-mismatch between the donor and the recipient, assays based on determining the frequency of sex-chromosomes may be used.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lamb, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD would only be shared following publication of the study.